CLINICAL TRIAL: NCT04780347
Title: A Phase II, Single-center, Randomized Study of Albumin-bound Paclitaxel Combination With Capecitabine Versus Capecitabine Monotherapy in Paclitaxel/Docetaxel-resistant Advanced Breast Cancer
Brief Title: Albumin-bound Paclitaxel Combination With Capecitabine Versus Capecitabine Monotherapy in Paclitaxel/Docetaxel-resistant Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Chief physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YBCSG-21-03
Record Dates: First submitted 2021-02-28; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Albumin-bound paclitaxel; paclitaxel/docetaxel-resistant
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin-bound paclitaxel plus capecitabine (Experimental): Albumin-bound paclitaxel combined with capecitabine
  Interventions: Drug: Albumin-bound paclitaxel plus capecitabine
- Capecitabine (Active Comparator): Capecitabine
  Interventions: Drug: capecitabine

INTERVENTIONS:
Drug: Albumin-bound paclitaxel plus capecitabine — Albumin-bound paclitaxel plus capecitabine: Albumin-bound paclitaxel 260mg/m2, IV , D1, q3w； capecitabine 1000 mg/m2, PO，bid, D1-14,q3w.
  Arms: Albumin-bound paclitaxel plus capecitabine
Drug: capecitabine — capecitabine: capecitabine 1000 mg/m2, PO，bid, D1-14,q3w.
  Arms: Capecitabine

SUMMARY:
Albumin-bound Paclitaxel Combination With Capecitabine Versus Capecitabine Monotherapy in Paclitaxel/Docetaxel-resistant Advanced Breast Cancer

DETAILED DESCRIPTION:
A Phase II, single-center, randomized study of albumin-bound paclitaxel combination with capecitabine versus capecitabine monotherapy in paclitaxel/docetaxel-resistant advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Females with age between 18 and 70 years old
2. Histological proven unresectable recurrent or advanced breast cancer
3. Negative for human epithelial receptor-2 (HER2) by immunohistochemistry. A negative Her2 gene amplification should be verified by FISH test for those patients with Her2 (2+). For those with Her2 (1+), FISH test might be considered by the investigator.
4. Patients who developed disease progression within 12 months of previous paclitaxel-containing chemotherapy regimens.
5. At least one measurable disease according to the response evaluation criteria in solid tumor (RECIST 1.1)
6. Performance status no more than 1
7. All patients enrolled are required to have adequate hematologic, hepatic, and renal function
8. Life expectancy longer than 12 weeks
9. No serious medical history of heart, lung, liver and kidney
10. Be able to understand the study procedures and sign informed consent.
11. Patients with good compliance.

Exclusion Criteria:

1. Pregnant or lactating women (female patients of child-bearing potential must have a negative serum pregnancy test within 14 days before the first day of drug dosing, or, if positive, a pregnancy should be ruled out by ultrasound)
2. Women of child-bearing potential, unwilling to use adequate contraceptive protection during the process of the study
3. Treatment with radiotherapy at the axial skeleton within 4 weeks before the first treatment or has not recovered from all toxicities of previous radiotherapy
4. Treatment with an investigational product within 4 weeks before the first treatment
5. Patients with symptomatic central nervous system metastases are not permitted, except for those with stable and asymptomatic brain metastases who have completed cranial irradiation, and have at least one measurable lesion outside the brain. Radiotherapy should be completed within 4 weeks prior to the registration
6. Other active malignancies (including other hematologic malignancies) or other malignancies within the last 5 years, except for cured nonmelanoma skin cancer or cervical intraepithelial neoplasia.
7. Patients having a history of clinically significant cardiovascular, hepatic, respiratory or renal diseases, clinically significant hematological and endocrinal abnormalities, clinically significant neurological or psychiatric conditions
8. Uncontrolled serious infection

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-02-25 (Estimated)

PRIMARY OUTCOMES:
PFS | approximately 6 weeks
  Progression Free Survival

SECONDARY OUTCOMES:
ORR | approximately 6 weeks
  Objective Response Rate
OS | Up to approximately 30 months
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided